CLINICAL TRIAL: NCT02750878
Title: A Randomized Controlled Trial of the Consent Process for Patients Undergoing Trans-obturator Tape Slings.
Brief Title: Surgical Consent Process for Trans-obturator Tape Slings.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Urogynecology Associates (Other)
Responsible Party: Principal Investigator, Eman Elkadry, M.D., MD, Fellowship Director, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 034-2015
Record Dates: First submitted 2016-04-14; First posted 2016-04-26 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urinary Incontinence, Stress [C13.351.968.934.814.500]
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Participants will receive only the standard verbal TOT surgical consent counseling.
- Intervention group (Other): Participants will receive the standard verbal TOT surgical consent counseling plus a handout describing their surgical intervention
  Interventions: Other: Informational Handout

INTERVENTIONS:
Other: Informational Handout
  Arms: Intervention group

SUMMARY:
The purpose of this study is to determine if addition of a handout to the standard consent process for the trans-obturator tape (TOT) mid-urethral sling procedure will improve patients' understanding, recall and satisfaction with their procedure. The information provided in the handout will include the procedure details, the accompanying risks and benefits, as well as the expectations and alternatives to the TOT procedure. The aim of the investigators is to improve and standardize the current process for surgical consent for patients undergoing a mid-urethral sling procedure, specifically the TOT. The investigators hypothesize that addition of a handout will improve patient's preoperative comprehension by an absolute value of 10% compared to the standard consent process. The investigators further hypothesize that the handout will improve patient satisfaction and recall of the surgical procedure details post operatively.

DETAILED DESCRIPTION:
This is a randomized controlled trial investigating whether adding an informational handout to the standard surgical consent will improve patient understanding, recall and satisfaction with their surgery. The primary outcome will be the patient's knowledge of her surgical details immediately before surgery. The secondary outcomes will be the patient's satisfaction, regret scale and the patient's postoperative knowledge of her surgery details.

A member of the research team will recruit eligible patients at their preoperative clinic visit during the signing of consent for their TOT surgery. Verbal counseling for the TOT surgical consent is the current standard of practice in the investigator's office. After the patient is counseled in the usual fashion and signs the consent for her planned TOT surgery, the patient will be offered participation in the study.

Eligible patients will be consented verbally by the investigators. After enrollment, patients will be randomized using a computer-generated block randomization scheme to allocate participants in a 1:1 ratio; randomization will be stratified by provider.

Participants will be randomized to one of two study arms:

1. Control Group: Participants will receive only the standard verbal TOT surgical consent counseling described above.
2. Intervention Group: Participants will receive the standard verbal TOT surgical consent counseling plus a handout describing their surgical intervention.

All participants will be asked to complete a baseline questionnaire at the enrollment visit. Participants randomized to the control group will be finished with this initial study visit after completing the baseline questionnaire. Participants randomized to the intervention arm will be given a handout describing the TOT procedure, risks and benefits, post-operative recovery and alternative treatment options, as discussed in the verbal surgical consent. The patient will be asked to read the handout and will then be given the handout to take home. The provider will answer any questions the patient has after reviewing the handout.

The next study encounter will occur in the preoperative area immediately prior to surgery. At this time all participants will be asked to complete a second questionnaire with questions similar to those in the baseline questionnaire.

The final study encounter will occur at the post-operative visit that occurs approximately six weeks after surgery. At this visit all participants will be asked to complete a final questionnaire. This questionnaire will be the same as the one administered immediately before surgery. All participants will also be asked to complete an additional questionnaire asking about satisfaction, regret and surgical experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ≥age 18
* Consented for TOT mid-urethral sling
* Able to read and understand English

Exclusion Criteria:

* History of surgical treatment for stress urinary incontinence using mid-urethral slings.
* Patients undergoing concomitant Trans-Obturator Post-Anal Sling (TOPAS) surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
A knowledge questionnaire at the pre-operative holding area to measure the patients' knowledge regarding their Trans Obturator Tape surgery. The percentage of correct answers will be reported and analyzed. | On the day of Trans Obturator Tape surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Auburn Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No